CLINICAL TRIAL: NCT00173979
Title: Tendon Mechanical Properties and Morphological Characteristics of Human Muscle
Brief Title: Tendon Mechanical Properties and Morphological Characteristics of Human Bicep and Tricep Muscles: An In Vivo Ultrasonographical Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700520
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2007-06-06 (Estimated); Status verified 2005-06

CONDITIONS: Healthy
Keywords: muscle; tendon

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
This current study tests whether the load-displacement and stress-strain characteristics of human bicep and tricep muscles and tendons change during graded maximal voluntary elbow extension and flexion exercises.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Age range from 18-35 years

Exclusion Criteria:

* History of shoulder/elbow which needs medical treatment or surgery

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Hsing-Kuo Wang, PhD, Study Director — School and Graduate Institute of Physical Therapy, NTU
Locations (1):
- School and Graduate Institute of Physical Therapy, NTU, Taiwan, Taipei, Taiwan